CLINICAL TRIAL: NCT04539327
Title: Analysis of the Clinical Experience With Rucaparib in the Rucaparib Access Program (RAP) in Spain - A GEICO Study
Status: Completed | Type: Observational
Sponsor: Grupo Español de Investigación en Cáncer de Ovario (Other)
Collaborators: Clovis Oncology, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: GEICO 87-R
Record Dates: First submitted 2020-08-10; First posted 2020-09-07 (Actual); Last update posted 2022-09-23 (Actual); Status verified 2022-09

CONDITIONS: Epithelial Ovarian Cancer; Fallopian Tube Cancer; Primary Peritoneal Cancer
Keywords: Rucaparib
MeSH Terms: conditions — Carcinoma, Ovarian Epithelial; Fallopian Tube Neoplasms | interventions — rucaparib

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Drug: Rucaparib — Participating local sites (GEICO-associated hospitals with expertise in gynecological cancer management) will enter clinical data of those patients who have previously participated in the rucaparib access program (RAP) in Spain and have given their consent.

SUMMARY:
The study consists of a retrospective observational, multicenter study in which the fundamental exposure factor being investigated is a drug (rucaparib).

A clinical database will be built including clinical data in three scenarios of rucaparib treatment: (1) platinum-sensitive BRCA-mutated patients after progression, (2) maintenance therapy in patients after a platinum-sensitive relapse in response, and (3) treatment therapy in BRCA-mutated patients who are currently platinum-resistant.

The specific objectives of the study are:

* To describe patient characteristics/medical history, safety, efficacy, and dosing of on-label treatment with rucaparib in real-world patients (real-world data).
* To describe patient characteristics/medical history, safety, efficacy, and dosing of all patients treated with rucaparib (including patients with on-label treatment and others) in real-world patients (real-world data).
* To show that data obtained in clinical trials could be reproduced in non-screened patients.

ELIGIBILITY:
Inclusion Criteria:

1. Written informed consent must be signed by all patients participating in the study who can be interviewed in the hospital (accessible, alive patients). Informed consent may not be required from unaccessible patients (dead, lost, etc.) according to ethics committee permissions and applicable law for retrospective studies in Spain.
2. Histological diagnosis of high-grade epithelial ovarian, fallopian tube, or primary peritoneal cancer treated in the context of rucaparib access program (RAP) in Spain.
3. Adult women (18 years or more at the time of diagnosis).

Exclusion Criteria:

1. Patients without medical record available (lost, empty or unretrievable clinical information).

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult (18 years or more) women diagnosed with high-grade epithelial ovarian, fallopian tube, or primary peritoneal cancer
Sampling Method: Non-Probability Sample
Enrollment: 52 (Actual)
Dates: Start 2020-07-29 (Actual); Primary Completion 2021-07-31 (Actual); Study Completion 2021-07-31 (Actual)

PRIMARY OUTCOMES:
Patient characteristics and medical history | Month 10-12
  Sex, age, mutational status (BRCA 1/2 [germline/somatic] and in other homologous recombination repair (HRR) genes), number of previous relapses, number of previous chemotherapy regimens, types of treatments received (chemotherapy, targeted therapies [bevacizumab, PARP inhibitors (PARPi)]), prior maintenance or with maintenance, treatment-free interval (platinum-based chemotherapy, non-platinum-based chemotherapy, targeted therapy).
Rucaparib safety data: Adverse Events | Month 10-12
  All rucaparib-related hematological and non-hematological, serious and non-serious adverse events (grade, start date, end date, action taken with rucaparib, outcome). In addition, adverse event treatments will be registered in the study database.
Rucaparib efficacy data | Month 10-12
Rucaparib dosing data | Month 10-12
Data reproducibility | Month 10-12
  In order to show that data obtained in clinical trials could be reproduced in non-screened patients, the outcomes will be discussed in the context of the results from ARIEL3 trial and the integrated analysis of Study 10 and ARIEL2.

CONTACTS AND LOCATIONS:
Overall Officials: Alfonso Yubero, Dr., Principal Investigator — Hospital Clínico Universitario Lozano Blesa
Locations (23):
- Spain (23):
  - Hospital Torrecárdenas, Almería, Andalusia
  - Hospital Universitario Virgen de la Victoria, Málaga, Andalusia
  - Hospital Universitario Virgen del Rocío, Seville, Andalusia
  - Hospital Universitario Nuestra Señora de Valme, Seville, Andalusia
  - Hospital General San Jorge, Huesca, Aragon
  - Hospital Clínico Universitario Lozano Blesa, Zaragoza, Aragon
  - Hospital Universitario Miguel Servet, Zaragoza, Aragon
  - Hospital Universitario Son Espases, Palma de Mallorca, Balearic Islands
  - Hospital del Mar, Barcelona, Catalonia
  - Hospital Clínic i Provincial, Barcelona, Catalonia
  - Complejo Hospitalario Universitario de Pontevedra, Pontevedra, Galicia
  - Hospital Universitario de Fuenlabrada, Fuenlabrada, Madrid
  - Hospital Universitario Infanta Sofía, San Sebastián de los Reyes, Madrid
  - Hospital Universitario de Araba Txagorritxu, Vitoria-Gasteiz, País Basco
  - Instituto Valenciano De Oncologia, Valencia, Valencia
  - Hospital Universitari i Politecnic La Fe, Valencia, Valencia
  - Hospital Público Lluis Alcanyis, Xàtiva, Valencia
  - Clínica Universidad de Navarra, Madrid
  - MD Anderson Cancer Center, Madrid
  - Hospital Clínico San Carlos, Madrid
  - Hospital Universitario Fundación Jiménez Díaz, Madrid
  - Hospital Universitario 12 Octubre, Madrid
  - Centro Integral Oncológico Clara Campal, Madrid